CLINICAL TRIAL: NCT00006373
Title: A Phase II Study of Intensive-Dose Topotecan, Ifosfamide/Mesna and Etoposide (Vepesid)(TIME) Followed by Autologous Stem Cell Rescue in High Risk Lymphoma
Brief Title: Combination Chemotherapy Followed by Bone Marrow or Peripheral Stem Cell Transplantation in Treating Patients With Non-Hodgkin's Lymphoma or Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-12246; MCC-12246; MCC-IRB-5670; SB-MCC-12246; NCI-G00-1865
Record Dates: First submitted 2000-10-04; First posted 2003-01-27 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Lymphoma
Keywords: stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult Burkitt lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Etoposide; Ifosfamide; Topotecan; Mesna

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TIME (Experimental): Topotecan, Ifosfamide, Mesna and Etoposide
  Interventions: Drug: etoposide; Drug: ifosfamide; Drug: topotecan hydrochloride; Procedure: autologous bone marrow transplantation; Drug: Mesna

INTERVENTIONS:
Drug: etoposide — Etoposide IV 500 mg/m2/day over 24 hours Days -5, -4, -3
  Other Names: vepesid(R); VP-16
Drug: ifosfamide — Ifosfamide 3,333 mg/m2/day IV over 2 hours (total dose 10,000 mg/m2)Days -8, -7, -6
  Other Names: Ifex(R)
Drug: topotecan hydrochloride — Topotecan 21.3 mg/m2/day (total dose 64 mg/m2 ) IV over 30 minutes Days -8, -7, -6
  Other Names: topotecan
Procedure: autologous bone marrow transplantation
Drug: Mesna — Mesna 1,111 mg/m2/dose IV over 30 minutes; 30 minutes before and 4 and 8 hours after ifosfamide (total dose 10,000 mg/m2) Days -8, -7, -6
  Other Names: Mesnex(R)

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell or bone marrow transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy followed by autologous bone marrow transplantation or peripheral stem cell transplantation in treating patients who have non-Hodgkin's lymphoma or Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of intensive high dose chemotherapy consisting of topotecan, ifosfamide, and etoposide followed by autologous bone marrow or peripheral blood stem cell transplantation in terms of response rate, progression free survival, and overall survival in patients with high risk non-Hodgkin's lymphoma or Hodgkin's lymphoma.
* Determine the pharmacokinetic profile of high dose topotecan and etoposide in these patients.
* Determine the pharmacodynamics and toxicity of this regimen in these patients.
* Determine the role of either an up or down regulation of DNA topoisomerase I or II amount and/or activity in terms of clinical response and toxicity in patients treated with this regimen.

OUTLINE: Patients receive intensive high dose chemotherapy consisting of ifosfamide IV over 2 hours followed by topotecan IV over 30 minutes on days -8 to -6 and etoposide IV continuously over 24 hours on days -5 to -3. Patients undergo autologous bone marrow or peripheral blood stem cell transplantation on day 0.

Patients are followed at 3, 6, and 12 months, annually until disease relapse, and then every 6 months until death.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-Hodgkin's lymphoma

  * No lymphoblastic lymphoma
  * Under 55 years of age:

    * Intermediate and high grade or aggressive disease that has relapsed and/or failed at least 2 salvage chemotherapy regimens OR
    * Failed to achieve complete response after first line induction chemotherapy and failed at least 1 salvage chemotherapy regimen
    * Low grade or indolent disease that has relapsed or failed to achieve complete response after first line induction chemotherapy and failed more than 2 salvage chemotherapy regimens
  * 55 years of age and over:

    * Intermediate and high grade or aggressive disease that has relapsed and/or failed to achieve complete response after first line induction chemotherapy
    * Low grade or indolent disease that has relapsed or failed to achieve complete response after first line induction chemotherapy OR
* Histologically confirmed Hodgkin's lymphoma

  * Under 55 years of age:

    * Received at least 2 prior salvage chemotherapy regimens
  * 55 years of age and over:

    * Stage III or IV disease that has relapsed or failed to achieve remission after combination induction chemotherapy
    * Prior primary radiotherapy allowed if relapse is high risk (e.g., recurrence in radiation field, B symptoms, or liver or bone marrow involvement)
* No active leptomeningeal involvement or severe symptomatic CNS disease

  * Prior CSF tumor involvement allowed if asymptomatic and no evidence of disease on lumbar puncture or no tumor involvement on MRI of the brain
* Solid tumors and brain metastases allowed

  * No evidence of disease by MRI and physical exam following optimal prior surgery and/or radiotherapy AND
  * At least 3 months since prior radiotherapy NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age:

* 18 to 64

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 2.0 mg/dL*
* SGOT or SGPT no greater than 2.5 times normal*
* No severe hepatic dysfunction NOTE: *Unless due to primary malignancy

Renal:

* Creatinine no greater than 2.0 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No severe cardiac dysfunction
* Ejection fraction at least 50% by MUGA scan
* Essential hypertension controlled by medication allowed

Pulmonary:

* DLCO at least 50% of normal OR
* No symptomatic obstructive or restrictive disease

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception
* No active infection
* HIV negative
* No insulin dependent diabetes mellitus
* No uncompensated major thyroid or adrenal dysfunction
* No significant skin breakdown from tumor or other disease
* No other prior malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* Prior doxorubicin or daunorubicin allowed if total dose no greater than 450 mg/m2
* No prior topotecan

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics

Surgery:

* See Disease Characteristics

Other:

* No concurrent nitroglycerin preparations for angina pectoris
* No concurrent antiarrhythmic drugs for major ventricular arrhythmias

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2000-02; Primary Completion 2006-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 3 years
  Progression-free survival as defined as the time from date of enrollment to the time of recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Steven C. Goldstein, MD, Study Chair — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States